CLINICAL TRIAL: NCT05103397
Title: High Dose Methylprednisolone Verses Low Dose in Correction of Congenital Acynotic Heart Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maha sadek El Derh, lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 171/2021
Record Dates: First submitted 2021-10-22; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Steroids; methyl prednisolonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose group (Active Comparator): low dose group. Group (A) (25 patients) patients will receive 10 mg/Kg methyl prednisolone after induction before separation to (CPB).
  Interventions: Drug: methyl prednisolone
- high dose group (Active Comparator): high dose group. Group (B) (25 patients) patients will receive 30 mg/Kg methyl prednisolone after induction before separation to (CPB).
  Interventions: Drug: Methyl Prednisolonate
- Placebo group (Placebo Comparator): placebo group. Group (C) (control group)(25 patients) patients will receive placebo in form of normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methyl prednisolone — Low dose group .Group (A) 10 mg/Kg methyl prednisolone will be received after induction and before separation to (CPB).
  Other Names: steroid
  Arms: low dose group
Drug: Methyl Prednisolonate — High dose group.Group (B) 30 mg/Kg will be received after induction and before separation (CPB)
  Other Names: steroid
  Arms: high dose group
Drug: Placebo — Placebo group.Group (C) (25 patients) patients will receive placebo in form of normal saline
  Arms: Placebo group

SUMMARY:
To compare the effect of low dose methylprednisolone versus high dose on inflammatory mediators' level and cardioprotective effect after CPB in correction of congenital acyanotic heart disease.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial, at Ain Shams University hospitals, Cardiovascular surgery hospital (cardiac surgery unit), Cairo, Egypt.

All patients' legal guardians will sign written informed consent before inclusion.

Randomization will be performed using a computer-generated randomization sequence.

Complete blood count, coagulation tests will be performed for all patients prior to the planned procedure. For all patients included in this study preoperative evaluation including a complete airway evaluation (mouth opening, mallampatii grading, thyromental distance, and evaluation of dentition) will be performed. Standard fasting guidelines will be checked. (Barash PG et al., 2006).

On patient's arrival to operating room, either inhalational induction by sevoflurane 4-6 % followed by an intravenous (IV) line insertion or IV induction by Ketamine 1-2 mg /kg and 0.01 mg / kg Atropine. Standard monitoring including electrocardiography (ECG), pulse oximetry (SpO2). Anesthesia technique: fentanyl 1-5 microgram/kg, will be given during mask preoxygenation with 100% oxygen, followed by non-depolarizing muscle relaxant (atracurium 0.5 mg /Kg) and then endotracheal intubation and capnography will be applied (Barash PG et al., 2006).

Femoral artery cannulation by 20 G Leader catheter cannula for invasive blood pressure (BP)measurement, triple lumen central line will be inserted in internal jugular vein (BRAUN) by ultrasound guided technique.

After achievement of anesthesia and full muscle relaxation and intubation of the airway, a blood sample ( 2 ml) will be taken to measure (IL6), Troponin I and blood glucose level. Skin incision will take place followed by median sternotomy. Heparin 300-500 IU/kg will be given before aortic cannulation to achieve ACT of 450-480 before starting CPB. Patients will then be divided into 3 groups:

Group (A) (25 patients) patients will receive 10 mg/Kg methyl prednisolone after induction before separation to (CPB). (Schroeder et al.,2003).

Group (B) (25 patients) patients will receive 30 mg/Kg methyl prednisolone after induction before separation to (CPB). (Keski-Nisula et al., 2013).

Group (C) (control group)(25 patients) patients will receive placebo in form of normal saline.

We will study the different doses of methylprednisolone as there is no standard dose confirmed in pediatric cardiac surgery. We will compare the low dose with high dose of this drug to decrease the different side effects of steroids, and we will detect the efficacy by measuring the inflammatory markers. In our institute the IL 6 is the only available marker to be measured.

The attending doctor will not give the drug, as another doctor not attending the surgery will give it. Both the attending doctor and intensivist will be blinded to the drug given.

After surgical correction of cardiac lesion and separation of cardiopulmonary bypass machine, support of the heart will be achieved and maintained by millirone 0.3-0.7 ug/Kg/min together with noradrenaline0.01-1 ug/Kg/min. Reversal of heparin by protamine sulphate 1:1 correction. Vital data, blood pressure and heart rate will be recorded every 10 minutes, the need or the dose of vasopressors needed will be recorded. After hemostasis and chest closure, patients will be transferred to ICU (Barash PG et al., 2006).

After admission to ICU, stabilization of patient, another blood sample of (2 ml) to measure (IL6) , troponin and random blood sugar will be taken, and a third sample will be withdrawn after 24 hours. Vital data will be recorded every 30 minutes till extubation. Time of extubation will be recorded. Complications like neurological events, occurrence of new arrhythmia, wound infection, ICU stay and mortality in the first seven days postoperative will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* We will include pediatric patients ( 1- 16) years old undergoing surgical correction for congenital acyanotic cardiac lesions needing cardiopulmonary bypass machine.

Exclusion Criteria:

* 1) Cyanotic heart disease. 2) Closed cardiac surgeries. 3) Previous cardiac surgery. 4) Patients suffering neurological illness. 5) Diabetics. 6) Emergency procedures. 7) Patients on preoperative steroid therapy. 8) Adult patients with congenital heart disease.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
assessment of Level of IL 6 after CPB time | 3 months
  comparing level of IL6 in different groups after CPB

SECONDARY OUTCOMES:
Less postoperative complications related to high doses of steroid represented as blood glucose level. | 3 months
  comparing Less postoperativecomplications related to high doses of steroid represented as blood glucose level.

CONTACTS AND LOCATIONS:
Locations (1):
- Samar mohammed, Cairo, Egypt